CLINICAL TRIAL: NCT05813067
Title: The Effects of JDS-HF3.0 on Vasomotor Symptoms in Menopausal Women: A Randomized, Double-Blinded, Placebo-Controlled Clinical Trial
Brief Title: Herbal Nutraceutical Supplementation on Vasomotor Symptoms in Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bonafide Health (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: B01-22-01-T0032
Record Dates: First submitted 2023-03-28; First posted 2023-04-14 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Vasomotor Symptoms; Postmenopausal Disorders
Keywords: Vasomotor Symptoms; Menopause; Women's Health

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled, parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Product: JDS-HF3.0 Capsules (Experimental): Dietary supplement containing a proprietary botanical blend with NK3R antagonistic activity
  Interventions: Dietary Supplement: JDS-HF 3.0
- Placebo Capsules (Placebo Comparator): Placebo capsule containing:
  * Microcrystalline cellulose
  * Silicon dioxide micronized
  * Magnesium stearate
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: JDS-HF 3.0 — Take 2 capsules once daily in the mornings with food
  Arms: Test Product: JDS-HF3.0 Capsules
Dietary Supplement: Placebo — Take 2 capsules once daily in the mornings with food
  Arms: Placebo Capsules

SUMMARY:
The role of nutrition is recognized as a vital component to healthy aging throughout menopause. The goal of this study is to evaluate a dietary supplement for its safety and effects on vasomotor symptoms in menopausal women.

DETAILED DESCRIPTION:
Menopause is characterized by the cessation of menstruation for 12 consecutive months. It is a natural phase in which a women's menstrual cycles permanently cease, with the transition often beginning around 50 years of age or older. Menopausal women often experience changes in vaginal health and sexuality, loss of bladder control, changes in mood, decreased sleep quality, changes in body composition, and vasomotor symptoms (VMS, including hot flashes and night sweats).

VMS can have a negative impact on quality of life by disrupting both sleep and mood. Some management strategies for VMS include hypnosis, and supplementation of vitamin E, black cohosh, and phytoestrogens. However, hormone replacement therapy still remains the most common and effective treatment. Hormone replacement therapy, using estrogen or estrogen-progestin containing products, reduces the frequency and severity of hot flashes by 75-79%. Although hormone replacement therapy is generally well tolerated, it has been linked to an increased risk of breast cancer. Due to this concern it is recommended to use hormone replacement therapy for the shortest duration and lowest dose possible. There is a need for alternative options to help manage VMS in menopausal women, and dietary supplements may fill this role.

The test product (TP) for this study is a dietary supplement containing a proprietary botanical blend containing polyphenols and flavonoids. These herbal ingredients have been previously investigated for various properties, which demonstrate the opportunity to support the quality of life of menopausal women experiencing VMS by improving sleep and mood.

This randomized, double-blind, placebo-controlled, parallel study will be conducted to evaluate the TP for its impacts on healthy menopausal women with VMS.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy menopausal women who are 40 to 65 years of age (inclusive).
2. Last menstrual period has occurred at least 6 months prior to screening.
3. MRS score ≥2 at screening and at baseline.
4. Have self-reported menopausal symptoms for the past 6 months.
5. Have self-reported at least five moderate to severe hot flashes per day (including night sweats), on average for 7 days
6. Have a body mass index (BMI) between 18.5 to 34.9 kg/m2 (inclusive).
7. In good general health (no active or uncontrolled diseases or conditions) and able to consume the study product.
8. Have normal vital signs or acceptable to the investigator vital signs (blood pressure and heart rate) at screening.
9. Agree to refrain from treatments for hot flashes and other symptoms of menopause.
10. Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures.

Exclusion Criteria:

1. Individuals who are lactating, pregnant or planning to become pregnant during the study.
2. Induced menopause through surgery such as bilateral oophorectomy or salpingo-oophorectomy, chemotherapy, radiation, or drugs.
3. Individuals who have had a partial or total hysterectomy.
4. Use of any treatment for menopausal symptoms or other concomitant treatments listed under the "concomitant therapies" section of the protocol
5. Have a known sensitivity, intolerability, or allergy to any of the study products or their excipients.
6. Received a vaccine for COVID-19 in the two weeks prior to screening or during the study period, current COVID-19 infections, or currently have the post COVID-19 condition as defined by World Health Organization (WHO) (i.e., individuals with a history of probable or confirmed SARS-CoV-2 infection, usually three months from the onset of COVID-19 with symptoms that last for at least two months and cannot be explained by an alternative diagnosis).
7. Have a positive medical history of heart disease, renal disease, hepatic impairment, or active systemic infection (e.g., lyme disease, TB, HIV).
8. Have uncontrolled high blood pressure (≥160 mmHg systolic or ≥100 mmHg diastolic) or thyroid disease, defined as not taking a stable dose of medication on the current regimen for a minimum of three months.
9. Have diabetes (Type I or Type II).
10. History of cancer (except localized skin cancer without metastases) within five (5) years prior to screening. Note: all women with breast cancer (active or any history) will be excluded.
11. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the potential subject at risk because of participation in the study, or influence the results or the potential subject's ability to participate in the study.
12. History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs (i.e., Crohn's disease, short bowel, acute or chronic pancreatitis or pancreatic insufficiency).
13. Active vaginal infections/abnormalities (e.g., active urinary tract infection (UTI), genital hemorrhage of unknown origin, pelvic inflammatory disease (PID)). Note: screened participants with infections would be eligible to participate four weeks after completing their treatment (wash-out period).
14. Participant has an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g., dysphagia) and digestion (e.g., known intestinal malabsorption, celiac disease, inflammatory bowel disease, chronic pancreatitis, steatorrhea).
15. Major surgery in three months prior to screening or planned major surgery during the study.
16. History of a surgical procedure for the treatment of obesity (e.g., gastric bypass, gastric banding).
17. History of alcohol or substance abuse.
18. Receipt or use of test product(s) in another research study within 28 days prior to the baseline visit (Day 1), or longer if the previous test product is deemed by the investigator to have lasting effects that might influence the eligibility criteria or outcomes of current study.
19. Use of any vaginal medications, rinses, moisturizers, cooling devices, cooling mattresses, cooling sprays, or patches purposed for hot flash control (i.e., V-cool patch, estrogen cream, etc.) one week before and during study.
20. Current or previous smoker in the last 3 years.
21. Any other active or unstable medical conditions or use of medications/supplements/ therapies that, in the opinion of the investigator, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 74 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
To determine the effects of the Test Product (TP) compared to placebo on hot flash symptoms as determined by the Hot Flash Related Daily Interference Scale (HFRDIS). | 12 weeks
  Change from baseline for the number and severity of hot flashes measured by HFRDIS scores.
  The HFRDIS has a scoring range of 0-100, with higher values indicating worse symptoms.

SECONDARY OUTCOMES:
To determine the effect of the TP compared to the placebo on overall menopausal symptoms as determined by the Greene Climacteric Scale (GCS). | 12 weeks
  Change from baseline in GCS scores.
  The GCS has 3 sub-domains for scoring. The psychological sub-domain has a scoring range from 0-33, the physical sub-domain has a scoring range from 0-21, and the vasomotor sub-domain has a scoring range from 0-6. Higher values indicate worse symptoms in all 3 sub-domains.
To determine the effect of the TP compared to the placebo on overall menopausal symptoms as determined by the Menopausal Rating Scale (MRS). | 12 weeks
  Change from baseline in MRS scores.
  The MRS has a scoring range of 0-44, with higher values indicating worse symptoms.
To determine the effect of the TP compared to the placebo on sleep quality as determined by the Pittsburgh Sleep Quality Index (PSQI). | 12 weeks
  Change from baseline in PSQI scores.
  The PSQI has a scoring range of 0-21, with higher values indicating worse symptoms.
To determine the effect of the TP compared to the placebo on quality of life as determined by the Menopause-Specific Quality of Life (MENQOL) questionnaire. | 12 weeks
  Change from baseline in MENQOL scores.
  The MRS has a scoring range of 0-174, with higher values indicating worse symptoms.

OTHER OUTCOMES:
To assess the safety and tolerability of the TP compared to the placebo in healthy participants. | 12 weeks
  Reports of adverse events (AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Samuel N Lederman, MD, Principal Investigator — Altus Research
Locations (3):
- United States (3):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Altus Research, Lake Worth, Florida
  - Rosemark WomenCare, Idaho Falls, Idaho

IPD SHARING:
Plan to Share IPD: No